CLINICAL TRIAL: NCT04649086
Title: Muscular Rehabilitation by Eccentric Exercise After Severe COVID-19 Infection: Research Protocol for Randomized Controlled Trial (CovExc)
Brief Title: Muscular Rehabilitation by Eccentric Exercise After Severe COVID-19 Infection
Acronym: CovExc
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Stop premature due to futility
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: GIRCI Auvergne Rhône-Alpes (Unknown); Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PHRCI 2020 COSTE (CovExc); 2020-A01201-38 (Other: ANSM)
Record Dates: First submitted 2020-09-29; First posted 2020-12-02 (Actual); Last update posted 2024-02-15 (Actual); Status verified 2021-05

CONDITIONS: Covid19; Sarcopenia; Muscle Weakness
Keywords: Covid19; Sarcopenia; Muscle Weakness; Eccentric exercises; Rehabilitation
MeSH Terms: conditions — COVID-19; Sarcopenia; Muscle Weakness

STUDY DESIGN:
Intervention Model Description: All included participants will be randomly assigned (1:1) using the REDCap software, , at the experimental group or the control group.
  Participants will perform 24 exercise sessions on cycloergometer (3 sessions/week, 8 weeks).
  The experimental group (eccentric) will perform 5 habituation sessions: the initial power of the exercise will be set to 10 Watts and then increased by 10% each session, depending on the muscle tolerance. The training power must correspond to 3 times that of the control group to obtain a similar metabolic stimulation.
  The control group (concentric) will perform exercise training at an intensity of 60% of the reserve heart rate determined during an initial cardiorespiratory test.
Masking Description: Evaluations will be carried out with blinding by investigators different from those involved in the exercise training sessions. Patients will be blinded to the training mode hypothesis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Eccentric group (Experimental): The experimental group (eccentric) will perform 5 habituation sessions: the initial power of the exercise will be set to 10 Watts and then increased by 10% each session, depending on the muscle tolerance. The training power must correspond to 3 times that of the control group to obtain a similar metabolic stimulation and will be adapted according to the pain felt at the end of the session.
  Interventions: Other: Rehabilitation by Eccentric exercises
- Concentric group (Active Comparator): The control group (concentric) will perform exercise training at an intensity of 60% of the reserve heart rate determined during an initial cardiorespiratory test. The power will be adjusted weekly to stay within the target heart rate range.
  Interventions: Other: Rehabilitation by Concentric exercises

INTERVENTIONS:
Other: Rehabilitation by Eccentric exercises — Participants will perform 24 exercises sessions (30 minutes) with cycloergometer in eccentric mode (while resisting against self-paced pedaling), inducing a greater muscular hypertrophy as compared with concentric mode, the mechanical stimulation being 3 to 4 times greater at the same level metabolic stimulation.
  Arms: Eccentric group
Other: Rehabilitation by Concentric exercises — The control group (concentric) will perform exercise training at an intensity of 60% of the reserve heart rate determined during an initial cardiorespiratory test. The power will be adjusted weekly to stay within the target heart rate range.
  Arms: Concentric group

SUMMARY:
With the COVID-19 pandemic, the number of patients to be treated in rehabilitation increased .

Hospitalization for severe infection can induce muscular atrophy and muscular dysfunction that persists for several months and rehabilitation capacities may be exceeded.

Exercises in eccentric mode could be performed, inducing greater muscular hypertrophy, muscle strength, power and speed than concentric exercises.

The goal of this study was to compare functional recovery at 2 months after a training program in eccentric and concentric mode after severe COVID-19.

An effective rehabilitation could help reduce costs and duration of care.

DETAILED DESCRIPTION:
This is a prospective, open, controlled randomized study (2 x 60 individuals) performed in 3 centers. Participants will perform 24 exercise sessions on cycloergometer (3 sessions/week, 8 weeks). The experimental group (eccentric) will perform 5 habituation sessions: the initial power of the exercise will be set to 10 Watts and then increased by 10% each session, depending on the muscle tolerance. The training power must correspond to 3 times that of the control group to obtain a similar metabolic stimulation. The control group (concentric) will perform exercise training at an intensity of 60% of the reserve heart rate determined during an initial cardiorespiratory test. The primary outcome will be the change in distance covered during the 6-min walk test between the initial assessment and month 2. Secondary outcomes will include study of sarcopenia, muscle strength, general and muscular fatigue, quality of life, blood metabolomic data, ex vitro data for mitochondrial and histo-biochemical functionality from muscle biopsies of the Vastus Lateralis.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, 18 to 80 years old
* Diagnosed for SARS-CoV-2 infection (COVID-19) requiring a rehabilitation program at least 1 month after the hospitalization
* Autonomy in daily life activities 1 month after diagnosis
* Able to walk for 6 min (discontinuous walking possible)
* Giving informed written consent to participate in the study
* Health insurance coverage

Exclusion Criteria:

* Cardiovascular or respiratory contraindication to the rehabilitation program
* Difficulty to perform an eccentric exercise on a seated ergometer
* Pregnant or breastfeeding
* Under guardianship, curatorship or deprived of liberty
* Taking antivitamin K anticoagulation (muscle biopsy)
* Refusal to participate

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-06-05 (Actual); Primary Completion 2022-01-07 (Actual); Study Completion 2022-01-07 (Actual)

PRIMARY OUTCOMES:
Functional walking capacity | Day 0, Month 1, Month 2 and Month 6
  Average change from baseline walking capacity measured by the 6-minutes walk test (6MWT), expressed in meters. All patients will be asked to cover the longest distance over a 30-meters distance in 6 min with or without stopping and with standardized verbal encouragements according to standard recommendations; to take into account a learning effect, the test will be performed twice, with the longer distance retained, expressed in meters. To prevent adverse effect, pulsed oxygen saturation (% of pSO²) and heart rate (heartbeat per minute) will be monitored continuously throughout the test by using a digital oximeter.

SECONDARY OUTCOMES:
Evaluating of lower extremity functioning by Short Physical Performance Battery (SPPB) score | Day 0, Month 2 and Month 6
  this test consists of assessing balance in a standing position, lifting from a chair (5 stand to-sit repetitions) and measuring 4-m walking speed (20). The patient walks 4 m at a normal and comfortable speed. The "test zone" (4 m) is preceded by an "acceleration zone" (1 m) and is followed by a "deceleration zone" (1 m). The assessor starts and stops the timing when the subject's foot meets the ground when entering and leaving the "test area", respectively.
Evaluating the maximum muscle strength of the quadriceps by Quadriceps Isometric Maximum Strength (QIMS) test | Day 0, Month 2
  maximum muscle strength of the quadriceps, on the dominant limb, will be measured on a bench: - Strength during isometric contraction (at 90° knee flexion) - Standardized position with the arms crossed on the chest, the absence of back support during the measurement and the maintenance of the hips and the contralateral leg to avoid any compensating movement Three reproducible measurements (±10%) will be taken at 1-min intervals, with the highest value retained.
Evaluating the fatigability of the quadriceps by Quadriceps Intermittent Fatigue (QIF) test | Day 0, Month 2
  this test consists of performing 10 knee extensions at 10% QIMS, then gradually increasing the load (10% by 10%) until exhaustion (cannot perform the movement 2 consecutive times). The value retained is the last level (% QIMS) performed.
Evaluating the global fatigability by Modified Fatigue Impact Scale (MFIS) | Day 0, Month 2 and Month 6
  this scale explores cognitive (10 items), physical (9 items) and psychosocial (2 items) fatigue. The MFIS included 21 items with a total score ranging from 0 to 84 with higher scores indicating a greater impact of quality of life.
Evaluating functional capacities with EuroQol - 5 Dimensions (EQ-5D) questionnaire | Day 0, Month 2 and Month 6
  This questionnaire explores 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. The EQ-5D-5L included 5 items independently scored from 1 to 5 (higher scores indicating a greater impact)and a 0-100 visual analogic scale exploring general health (0 means the worst heath patient can imagine, 100 means the best health patient can imagine).
Evaluating the handgrip strength by standard handgrip strength test | Day 0, Month 2
  measurement is in 90° elbow flexion, wrist in neutral position. Three reproducible measurements (± 10%) will be taken at 1-min intervals, with the highest value retained.
Metabolomic Profile | Day 0, Month 2 (post-training)
  Plasma metabolome profile assessed by variation of number of blood metabolites. Changes from baseline to post-training intervention in plasma metabolome profile will be compared between excentric and concentric exercise groups.
Cross sectional area measurement | Day 0, Month 2 (post-training)
  Biopsy from the Vastus lateralis will be performed and the variation of cross sectional area measurement of muscle fibers (µm2) will be analysed and compared between excentric and concentric exercise groups from baseline to post-training intervention.
Capillary to fibre ratio. | Day 0, Month 2 (post-training)
  Biopsy from the Vastus lateralis will be performed and the capillarization (variation of capillary to fiber ratio) will be analysed.
  Muscle adapations from baseline to post-training intervention will be compared between excentric and concentric exercise groups.
Satellite cell number | Day 0, Month 2 (post-training)
  Biopsy from the Vastus lateralis will be performed and the evolution of number of satellite cell per muscle fiber will be analysed and compared between excentric and concentric exercise groups from baseline to post-training intervention.
Neuromuscular activation | Day 0, Month 2 (post-training)
  Electrophsyiological stimulation of the quadriceps for the measurement of the neuromuscular activation before, during and after the QIF test. During this test, we measure maximal M-wave, contraction time and torque and the percentage of neuromuscular activation. Neuromuscular activation will be analysed and compared between excentric and concentric exercise groups from baseline to post-training intervention.
Quadriceps muscular Oxygen Tissue Saturation | Day 0, Month 2 (post-training)
  An infrared spectroscopy device is localized on the anterior part of the quadriceps. The device measures hemoglobin and desoxyhemoglobin concentration under the placement area. This measure is performed, before, during and after the QIF test. During this test, we measure the hemoglobin and desoxyhemoglobin concentration as well as the tissue saturation index.Quadriceps muscular Oxygen Tissue Saturation will be analysed and compared between excentric and concentric exercise groups from baseline to post-training intervention.
O2 uptake Efficiency during walk test | Day 0, Month 2 (post-training)
  A gaz exchange device records the O2 uptake during the 6 minutes walk test. The O2 uptake efficiency was defined as the volume of O2 per meter used by the participant.
  An infrared spectroscopy device is localized on the anterior part of the quadriceps. O2 uptake Efficiency during walk test will be analysed and compared between excentric and concentric exercise groups from baseline to post-training intervention.
Creatine Kinase (CPK) | Day 0
  A blood sample collection to measure the CPK concentration.
Creatine Kinase (CPK) | Day 7 (post-training)
  A blood sample collection to measure the CPK concentration.
Creatine Kinase (CPK) | Month 2 (post-training)
  A blood sample collection to measure the CPK concentration.
C-reactive protein (CRP) | Day 0
  A blood sample collection to measure CRP concentration.
C-reactive protein (CRP) | Day 7 (post-training)
  A blood sample collection to measure CRP concentration.
C-reactive protein (CRP) | Month 2 (post-training)
  A blood sample collection to measure CRP concentration.

CONTACTS AND LOCATIONS:
Overall Officials: Maxime GROLIER, MD, MSc, Principal Investigator — CHU de Clermont-Ferrand; Emmanuel COUDEYRE, MD, PhD, Study Director — CHU de Clermont-Ferrand
Locations (3):
- France (3):
  - CHU de Clermont-Ferrand, Clermont-Ferrand
  - CHU de Dijon, Dijon
  - CHU de Saint-Etienne, Saint-Etienne

REFERENCES:
- [Background] Zhang P, Li J, Liu H, Han N, Ju J, Kou Y, Chen L, Jiang M, Pan F, Zheng Y, Gao Z, Jiang B. Long-term bone and lung consequences associated with hospital-acquired severe acute respiratory syndrome: a 15-year follow-up from a prospective cohort study. Bone Res. 2020 Feb 14;8:8. doi: 10.1038/s41413-020-0084-5. eCollection 2020. PMID 32128276
- [Background] Puthucheary ZA, Rawal J, McPhail M, Connolly B, Ratnayake G, Chan P, Hopkinson NS, Phadke R, Dew T, Sidhu PS, Velloso C, Seymour J, Agley CC, Selby A, Limb M, Edwards LM, Smith K, Rowlerson A, Rennie MJ, Moxham J, Harridge SD, Hart N, Montgomery HE. Acute skeletal muscle wasting in critical illness. JAMA. 2013 Oct 16;310(15):1591-600. doi: 10.1001/jama.2013.278481. PMID 24108501
- [Background] Connolly B, Salisbury L, O'Neill B, Geneen L, Douiri A, Grocott MP, Hart N, Walsh TS, Blackwood B. Exercise rehabilitation following intensive care unit discharge for recovery from critical illness: executive summary of a Cochrane Collaboration systematic review. J Cachexia Sarcopenia Muscle. 2016 Dec;7(5):520-526. doi: 10.1002/jcsm.12146. Epub 2016 Sep 16. PMID 27891297
- [Background] van Zanten ARH, De Waele E, Wischmeyer PE. Nutrition therapy and critical illness: practical guidance for the ICU, post-ICU, and long-term convalescence phases. Crit Care. 2019 Nov 21;23(1):368. doi: 10.1186/s13054-019-2657-5. PMID 31752979
- [Background] Wu Y, Xu X, Chen Z, Duan J, Hashimoto K, Yang L, Liu C, Yang C. Nervous system involvement after infection with COVID-19 and other coronaviruses. Brain Behav Immun. 2020 Jul;87:18-22. doi: 10.1016/j.bbi.2020.03.031. Epub 2020 Mar 30. PMID 32240762
- [Background] Bailey P, Thomsen GE, Spuhler VJ, Blair R, Jewkes J, Bezdjian L, Veale K, Rodriquez L, Hopkins RO. Early activity is feasible and safe in respiratory failure patients. Crit Care Med. 2007 Jan;35(1):139-45. doi: 10.1097/01.CCM.0000251130.69568.87. PMID 17133183
- [Background] Needham DM. Mobilizing patients in the intensive care unit: improving neuromuscular weakness and physical function. JAMA. 2008 Oct 8;300(14):1685-90. doi: 10.1001/jama.300.14.1685. PMID 18840842